CLINICAL TRIAL: NCT00253500
Title: Prediction of Response or Resistance to Dose Intensified Pre-Operative Epirubicin Therapy of Operable Breast Cancer
Brief Title: Epirubicin in Treating Women Who Are Undergoing Surgery for Stage I, Stage II, or Stage III Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE3104
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage I breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pegfilgrastim; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Epirubicin (Experimental)
  Interventions: Biological: pegfilgrastim; Drug: epirubicin hydrochloride; Procedure: conventional surgery

INTERVENTIONS:
Biological: pegfilgrastim — 6 mg in a syringe
  Other Names: Neulasta
Drug: epirubicin hydrochloride — 120 MG q 2 weeks for 4 cycles
Procedure: conventional surgery — to remove small piece of cancer
  Other Names: Biopsy will involve a small surgical incision to remove a piece of the cancer.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as epirubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving epirubicin before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well epirubicin works in treating women who are undergoing surgery for stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the complete pathological and clinical response rate in women undergoing surgery for resectable stage I-III breast cancer treated with neoadjuvant dose-intensified epirubicin hydrochloride.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine the predictive value of HER2 gene amplification and topoisomerase II-alpha gene amplification or deletion for disease progression and pathological and clinical complete response in patients treated with this regimen.
* Correlate gene expression profiles with pathologic complete response, clinical complete response, less than complete response, and disease progression in patients treated with this regimen.

OUTLINE: Patients receive epirubicin hydrochloride IV on day 1 and pegfilgrastim subcutaneously on day 2. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity. Four weeks later, patients undergo partial mastectomy or simple mastectomy plus an axillary staging procedure.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer

  * Stage I, II, or III disease (T1, T2, or T4; N0-2; M0)

    * Resectable disease
* Unidimensionally measurable disease

  * Primary tumor ≥ 2 cm
* No known distant metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Sex

* Female

Menopausal status

* Not specified

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 3,500/mm^3
* Hemoglobin ≥ 8 g/dL
* Platelet count ≥ 100,000/mm^3
* No known untreated bleeding diathesis

Hepatic

* AST ≤ 2 times upper limits of normal
* Bilirubin ≤ 1.5 mg/dL

Renal

* Creatinine ≤ 1.5 mg/dL OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* LVEF ≥ 50% on echocardiogram, MUGA, or cardiac catheterization

Other

* Not pregnant or breastfeeding
* Fertile patients must use effective contraception
* Negative pregnancy test
* No concurrent illness that would preclude study treatment
* No known hypersensitivity to Escherichia coli-derived proteins, pegfilgrastim, filgrastim (G-CSF), or any other component of these products

PRIOR CONCURRENT THERAPY: Not specified

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2002-06; Primary Completion 2005-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Complete pathological response rate by tumor analysis after surgery | 4 weeks
  No evidence of microscopic invasive tumor at the primary tumor site in the surgical specimen.

SECONDARY OUTCOMES:
Complete clinical response rate by diagnostic mammogram at baseline and at 8 weeks | 4 weeks
  Bilateral (if both breasts are present) Mammograms (within 4 weeks of study entry)
Toxicity by physical exam and medical history every 14 days prior to surgery | 2-4 weeks
  A physical exam Physical examination with recording of tumor size, if palpable.
Predictive value of HER2 gene amplification and topoisomerase II-alpha gene amplification or deletions for pathologic complete response, clinical complete response or disease progression after surgery | 5 years
  Patients whose tumors are positive for estrogen receptor (>1% staining by immunohistochemistry) or progesterone receptor (institutional definition) should receive post-operative hormonal therapy for 5 years.
Gene expression after surgery | 5 years
  Patients whose tumors are positive for estrogen receptor (>1% staining by immunohistochemistry) or progesterone receptor (institutional definition) should receive post-operative hormonal therapy for 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: George T. Budd, MD, Study Chair — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://clinicaltrials.gov/ct2/results?term=case3104